CLINICAL TRIAL: NCT03948048
Title: Study on the Efficacy and Timing of Extracorporeal Membrane Oxygenation (ECMO) Therapy in Children With Refractory Septic
Brief Title: Study on the Efficacy and Timing of ECMO Therapy in Children With Refractory Septic Shock
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Children's Hospital (Other); Beijing Children's Hospital (Other); Zhengzhou Children's Hospital, China (Other); Chinese PLA General Hospital (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); Children's Hospital of Chongqing Medical University (Other); Shengjing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: fdpicu-03
Record Dates: First submitted 2019-05-10; First posted 2019-05-13 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Septic Shock; Extracorporeal Membrane Oxygenation Complication
Keywords: septic shock; children; ECMO; timing
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- septic shock: The critically ill children with septic shock (ss group)
- refractory septic shock with ECMO: The critically ill children with refractory septic shock with ECMO treatment
  Interventions: Device: ECMO
- refractory septic shock without ECMO: The critically ill children prediction model th refractory septic shock without ECMO treatment

INTERVENTIONS:
Device: ECMO — ECMO is used to intervene septic shock and refractory septic shock
  Groups: refractory septic shock with ECMO

SUMMARY:
Severe sepsis and septic shock remain the leading causes of child mortality worldwide. Sepsis is a complex process that ultimately leads to circulation disorders, organ perfusion abnormalities, capillary leakage, tissue hypoxia, and organ failure. The difficulty of clinical treatment is microcirculation and mitochondrial dysfunction in septic shock. Once shock enters the stage of microcirculation failure, conventional treatment is ineffective. ECMO can effectively support the circulatory system and provide good oxygen delivery, but there are many controversies in clinical treatment. 1) whether ECMO can effectively improve the clinical prognosis of children with septic shock; 2) appropriate timing for ECMO intervention; 3) which key clinical factors affect the effect of ECMO treatment. This study intends to adopt a multi-center, prospective, non-randomized controlled trial design, and the main research hypothesis is whether ECMO treatment can improve the success of discharge survival of children with septic shock.

DETAILED DESCRIPTION:
In this study, a variety of statistical analysis methods will be used to screen the clinical indicators and truncation values suitable for starting ECMO, and to construct a comprehensive prediction model, so as to determine the basis for the optimal timing of ECMO treatment in the future. The efficacy of ScVO2, lactic acid, and vasoactive inotrope score (VIS) on the ECMO treatment timing will also be evaluated. This study aims to evaluate and improve the clinical application of ECMO in the treatment of sepsis in children

ELIGIBILITY:
Inclusion Criteria:

• Children with septic shock and refractory septic shock admitted to the PICU of all the study centers

Exclusion Criteria:

* Fatal chromosomal abnormalities (e.g., trisomy 13 or 18)
* Uncontrolled bleeding
* Irreversible brain damage
* After allogeneic bone marrow transplantation
* Weight less than 2.5kg or severe malnutrition

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with septic shock and refractory septic shock admitted to the pediatric intensive care unit（PICU） of all the study centers
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 28 days
  The survival rate of children in 28 days after hospital discharge

SECONDARY OUTCOMES:
ECMO weaning rate | 48 hours
  The success of ECMO weaning is defined as the survival of patients after ECMO weaning for 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Guoping Lu, Doctor, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children'S Hosptial of Fuan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided